CLINICAL TRIAL: NCT04035356
Title: Safety and Performance of Aortic Valve Repair Using the HAART Aortic Annuloplasty Devices - A Registry Study
Brief Title: HAART Annuloplasty Device Valve Repair Registry
Status: Terminated | Type: Observational
Why Stopped: The study will be merged with another one.
Sponsor: Biostable Science & Engineering (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-01-045
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Aortic Valve Insufficiency; Aortic Aneurysm
Keywords: aortic valve repair; aortic valve annuloplasty
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- HAART 300: HAART 300 Aortic Annuloplasty Device
  Interventions: Device: Aortic valve repair
- HAART 200: HAART 200 Aortic Annuloplasty Device
  Interventions: Device: Aortic valve repair

INTERVENTIONS:
Device: Aortic valve repair — Use of a HAART Aortic Annuloplasty Device in patients undergoing aortic valve repair surgery

SUMMARY:
Multicenter US registry study to assess procedure success and long-term (10-year) performance of the HAART 200 and HAART 300 Aortic Annuloplasty Devices when used during aortic valve repair in a routine cardiovascular practice setting.

DETAILED DESCRIPTION:
The HAART Aortic Annuloplasty Devices are three-dimensional annuloplasty rings designed to be implanted intra-annularly in the aortic valve to correct annular dilatation and/or maintain annular geometry of the aortic valve in patients with trileaflet valve morphology (HAART 300) or bicuspid valve morphology (HAART 200) with moderate to severe aortic insufficiency who are undergoing aortic valve repair due to symptoms or as part of a repair for an aortic aneurysm.

The study is a multicenter registry study enrolling both retrospective and prospective participants. Investigators are cardiothoracic surgeons specializing in surgery of the aortic valve and aorta at facilities with suitable infrastructure to support collection of the registry study data. Patients who underwent or will undergo aortic valve repair using either the HAART 300 or HAART 200 Device will be enrolled. All patients known to have received the HAART 300 or HAART 200 Device at participating centers will be contacted and offered the opportunity to enroll in this registry study. Prospective participants will have evaluations prior to surgery, intraoperatively, immediately following surgery, at discharge (or within 90 days), and at 1, 3, 5, and 10 years. In addition to the follow-up clinic visits, phone contacts are scheduled at years 2,4,6, 7, 8, and 9 to maintain participant engagement as well as to ascertain if any safety events have taken place. Retrospective participants who have already received the HAART 300 or HAART 200 Device prior to study enrollment will undergo safety assessment at the time of enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* The patient underwent or is undergoing aortic valve repair using either the HAART 300 or HAART 200 Aortic Annuloplasty Device in accordance with the Instructions for Use.
* The patient has reviewed and signed the written informed consent form.
* The patient agrees to return for all follow-up evaluations for the duration of the study.

Exclusion Criteria:

* Retrospective patient that has undergone a subsequent aortic valve replacement procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent or will undergo aortic valve repair using either the HAART 300 or HAART 200 Device at participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Freedom from aortic valve reoperation | 10 years
  A reintervention for repair or replacement of the aortic valve will be considered failure for this outcome measure

OTHER OUTCOMES:
NYHA Functional Classification | 10 years
  New York Hospital Association (NYHA) class:
  * Class I: cardiac disease but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain.
  * Class II: cardiac disease resulting in slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  * Class III: cardiac disease resulting in marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain.
  * Class IV: cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Aortic valve regurgitation grade | 10 years
  The severity of aortic valve regurgitation expressed as the aortic regurgitation (AR) Grade (or Aortic insufficiency (AI) Grade). The grades are defined by the American Society of Echocardiography guidelines based on regurgitant volume (RVol), regurgitant fraction (RF), and effective regurgitant orifice area (EROA), and expressed as:
  0 (None/trace)
  I (Mild: RVol <30 mL, RF <30%, EROA <0.1 cm**2)
  II (Mild-Moderate: RVol 30-44 mL, RF 30-39%, EROA 0.1-0.19 cm**2)
  III (Moderate-Severe: RVol 45-59 mL, RF 40-49%, EROA 0.20.29 cm**2)
  IV (Severe: RVol ≥60 mL, RF ≥50%, EROA ≥0.3 cm**2).
Freedom from Cardiovascular Events | 10 years
  Occurrence of any of the following events will be considered failure on this outcome measure.
  * Cardiac-related death
  * Aortic valve reintervention/reoperation
  * Major bleeding event
  * Structural valve deterioration
  * Nonstructural dysfunction
  * Operated valve endocarditis
  * Valve thrombosis
  * New permanent pacemaker or defibrillator within 14 days after the valve intervention
  * Embolism
All cause mortality | 10 years
  Death due to any cause
Noncardiovascular serious adverse events | 10 years
  Adverse events not of cardiovascular nature that led to death, resulted in a life-threatening illness or injury, resulted in hospitalization, or resulted in persistent or significant disability/incapacity.

CONTACTS AND LOCATIONS:
Overall Officials: J. Scott Rankin, MD, Principal Investigator — West Virginia University Heart and Vascular Institute
Locations (5):
- United States (5):
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - West Virginia University Heart & Vascular institute, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mazzitelli D, Fischlein T, Rankin JS, Choi YH, Stamm C, Pfeiffer S, Pirk J, Detter C, Kroll J, Beyersdorf F, Griffin CD, Shrestha M, Nobauer C, Crooke PS, Schreiber C, Lange R. Geometric ring annuloplasty as an adjunct to aortic valve repair: clinical investigation of the HAART 300 device. Eur J Cardiothorac Surg. 2016 Mar;49(3):987-93. doi: 10.1093/ejcts/ezv234. Epub 2015 Jul 8. PMID 26156945
- [Background] Mazzitelli D, Pfeiffer S, Rankin JS, Fischlein T, Choi YH, Wahlers T, Nobauer C, Schreiber C, Lange R. A Regulated Trial of Bicuspid Aortic Valve Repair Supported by Geometric Ring Annuloplasty. Ann Thorac Surg. 2015 Jun;99(6):2010-6. doi: 10.1016/j.athoracsur.2015.01.050. Epub 2015 Apr 10. PMID 25865762
- [Background] Rankin JS, Mazzitelli D, Fischlein T, Choi YH, Pirk J, Pfeiffer S, Wei LM, Badhwar V. Geometric Ring Annuloplasty for Aortic Valve Repair During Aortic Aneurysm Surgery: Two-Year Clinical Trial Results. Innovations (Phila). 2018 Jul/Aug;13(4):248-253. doi: 10.1097/IMI.0000000000000539. PMID 30138245